CLINICAL TRIAL: NCT07064642
Title: A Retrospective Comparison Of The Effects Of Low-Flow And High-Flow Anesthesia On Hemodynamics, Neutrophil-To-Lymphocyte Ratio, And Postoperative Outcomes In Tympanoplasty And Myringoplasty Surgeries
Brief Title: NLR and Sevoflurane Use in Ear Surgeries: Flow Comparison
Acronym: ANFLUX
Status: Completed | Type: Observational
Sponsor: Eda KAZANÇ ÖZDEN (Other)
Responsible Party: Sponsor-Investigator, Eda KAZANÇ ÖZDEN, Resident Doctor in Anesthesiology, Sponsor-Investigator, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Other Study IDs: EKO-NLR-2025; 2023/122 (Other: Karadeniz Technical University Faculty of Medicine Ethics Committee)
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Tympanoplasty; Myringoplasty; Neutrophil-to-Lymphocyte Ratio; Low-flow Anesthesia; High-flow Anesthesia
Keywords: Anesthesia high-flow; Anesthesia low-flow; Neutrophil-lymphocyte ratio; Systemic inflammatory response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-flow anesthesia group: Low-flow anesthesia group 0.75 L/min :
  Patients who underwent tympanoplasty or myringoplasty under low-flow anesthesia technique. The anesthetic gas flow rate was maintained at low levels throughout the procedure to evaluate its effects on systemic inflammation and hemodynamics.
- High-flow anesthesia group: High-flow anesthesia group 3 L/min :
  Patients who underwent tympanoplasty or myringoplasty under high-flow anesthesia technique. The anesthetic gas flow rate was maintained at high levels throughout the procedure to compare its impact on inflammatory response and postoperative outcomes.

SUMMARY:
This retrospective study aims to compare the effects of low-flow and high-flow anesthesia techniques on intraoperative hemodynamics, neutrophil-to-lymphocyte ratio (NLR), and postoperative outcomes in patients undergoing tympanoplasty or myringoplasty. The data were collected from medical records of patients who underwent ear surgery between [September 1, 2022] and [April 1, 2023]. The study seeks to evaluate whether the choice of anesthetic flow rate has a significant impact on inflammatory response and recovery.

DETAILED DESCRIPTION:
This study investigates the influence of anesthetic gas flow rates on systemic inflammation and hemodynamic stability in middle ear surgeries. While low-flow anesthesia is associated with reduced environmental exposure and cost-effectiveness, its impact on inflammatory markers and recovery outcomes remains less clearly defined. The neutrophil-to-lymphocyte ratio (NLR) is used as a readily available, cost-effective biomarker of systemic inflammation. This study retrospectively analyzes perioperative data from patients who underwent tympanoplasty or myringoplasty, comparing NLR levels, intraoperative vital signs, and postoperative recovery parameters between low-flow and high-flow anesthesia groups. The results may contribute to optimizing anesthetic strategies in otologic surgeries, with emphasis on inflammation modulation and patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 75 years
* American Society of Anesthesiologists (ASA) physical status classification I to III
* Body Mass Index (BMI) between 18.5 and 29.9 kg/m²

Exclusion Criteria:

* Age below 18 or above 75 years
* Incomplete or missing clinical data
* BMI less than 18.5 kg/m² or greater than 29.9 kg/m²
* Presence of neurological disorders
* History of renal or hepatic failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study evaluated patients who underwent tympanoplasty or myringoplasty surgery at the operating rooms of Karadeniz Technical University Faculty of Medicine between September 1, 2022, and April 1, 2023. Participants were excluded based on the following criteria: age under 18 or over 75 years, incomplete clinical data, body mass index (BMI) <18.5 kg/m² or >29.9 kg/m², presence of neurological disorders, and a history of renal or hepatic failure. A total of 59 patients aged between 18 and 75 years, with ASA (American Society of Anesthesiologists) physical status scores of I-III and BMI values between 18.5 and 29.9 kg/m², were initially included in the study. Following the exclusion of nine patients with missing data, the final study population consisted of 50 individuals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Postoperative neutrophil-to-lymphocyte ratio (NLR) | Within 1 hour postoperatively (Day 0)
  The neutrophil-to-lymphocyte ratio measured from blood samples taken immediately after surgery to assess the systemic inflammatory response in patients undergoing tympanoplasty or myringoplasty with low-flow or high-flow anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University Faculty of Medicine Hospital, Trabzon, Trabzon, Turkey (Türkiye)